CLINICAL TRIAL: NCT02126020
Title: Topical Infliximab in Autoimmune Eyes With Keratoprosthesis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patients met eligibility criteria. The study has been closed.
Sponsor: James Chodosh, MD, MPH (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other); Fonds de recherche en ophtalmologie de l'Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, James Chodosh, MD, MPH, Associate Director of the Cornea and Refractive Surgery Service, Director of Boston Keratoprosthesis Clinical Programs, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEEI 13-110H; IND 122719 (Other: FDA)
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolysis (Lyell) Syndrome; Mucous Membrane Pemphigoid
Keywords: Keratoprosthesis; corneal melt; keratolysis; Tumor necrosis factor alpha; infliximab; matrix metalloproteinase
MeSH Terms: conditions — Stevens-Johnson Syndrome; Syndrome; Pemphigoid, Benign Mucous Membrane | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topical infliximab (Experimental): topical infliximab 10 mg/mL QID x 3 months followed by BID x 9 months
  Interventions: Drug: topical infliximab

INTERVENTIONS:
Drug: topical infliximab — topical infliximab administered QID for 3 months followed by BID for 9 months
  Other Names: Remicade

SUMMARY:
The Boston Keratoprosthesis type I (KPro) is a prosthetic cornea used to treat several causes of corneal blindness. Some categories of patients, including those with auto-immune diseases such as Stevens-Johnson syndrome, toxic epidermal necrolysis syndrome and mucous membrane pemphigoid, have a higher risk of failure for the KPro. Because of chronic inflammation, the cornea supporting the KPro may melt, leading to a higher risk of infection, loss of the KPro and loss of the eye.

Infliximab is an antibody against tumor necrosis factor alpha and is used intravenously to control inflammation in several diseases. It has been used in some cases of corneal melting with significant success.

This study's hypothesis is that infliximab can be successfully used as an eye drop (instead of the usual administration through veins) and that its regular use may prevent melt in eyes with a Boston Keratoprosthesis type I and underlying auto-immune disease.

DETAILED DESCRIPTION:
This is an unmasked, prospective, multicenter clinical trial of four patients that are candidates for a Boston Keratoprosthesis or have had prior KPro surgery and have a diagnosis of Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis syndrome (TENS) or mucous membrane pemphigoid (MMP). Only one eye per patient will be considered for inclusion.

This is a phase I/II study to evaluate the safety and tolerance of topical infliximab 10 mg/mL eye drops. Research subjects will be required to administer infliximab eye drops four times per day for three months followed by twice daily administration for nine months. The subjects will be monitored while on the study medication as well as for one year following discontinuation of the drug. The total study duration for each patient will be two years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Able to provide informed consent
* Underlying diagnosis of SJS, TENS, or MMP
* Implantation of a Boston KPro type I
* Able to administer eye medications or have a care giver able and willing to do same
* Negative tuberculosis screening

Exclusion Criteria:

* Active or recurrent ocular or systemic infection

  * Chest radiography, QuantiFERON-TB Gold or purified protein derivative (PPD) evidence of active or latent tuberculosis infection
  * Indeterminate initial and repeat QuantiFERON-TB Gold results
  * History of Bacille Calmette-Guerin (BCG) vaccination within twelve months of screening
  * History of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening
  * Chest radiograph within three months prior to the first administration of the study drug that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis.
  * History of a nontuberculous mycobacterial infection or opportunistic infection (e.g. cytomegalovirus, pneumocystosis, aspergillosis) within six months prior to screening
  * history of hepatitis B virus
  * Methicillin resistant Staphylococcus aureus (MRSA) or vancomycin resistant enterococcus (VRE) infection
* Malignancy diagnosed in the last five years
* Demyelinating disease
* History or current diagnosis of diabetes mellitus (controlled and uncontrolled)
* Heart failure (New York Heart Association class III or IV)
* Pregnancy or breast-feeding
* Scheduled to receive a live vaccine at any time point during study participation
* Allergy to infliximab or any of the compounds in its topical formulation or any chemically-related medication
* Prior or current use of systemic anti-tumor necrosis alpha-α medications or currently receiving treatments of Kineret (Anakinra)
* KPro designs with less than 16 holes in the back plate (to avoid the confounder of corneal nutrition)
* Inability to comply with the instillation of additional drops
* Unable to attend postoperative visits or administer medications, or no care giver available and willing to assist with same

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Estimated)

PRIMARY OUTCOMES:
Tolerability | 1 year
  Percentage of patients finishing 12 months of topical infliximab use
Adverse events | 2 years
  Number and type of adverse events
rate of corneal melting | 2 years
  rate of corneal melting or ulceration during infliximab prophylaxis (12 months) and after the drug is stopped (following 12 months)
KPro retention | 2 years
  Percentage of retained KPros at 2 years

SECONDARY OUTCOMES:
Visual acuity | 2 years
Ocular surface symptoms | 2 years
  Ocular surface symptoms as assessed by ocular surface disease index score
Ocular surface inflammation | 2 years
  Ocular surface inflammation using slit-lamp photographs and the ocular redness index (ORI)
tear matrix metalloproteinase (MMP) | 2 years
  Levels and activity of MMPs, myeloperoxidase and tissue inhibitor of MMP-1
graft thickness | 2 years
  Corneal carrier graft thickness as measured by anterior segment optical coherence tomography before, during and after treatment with infliximab

CONTACTS AND LOCATIONS:
Overall Officials: James Chodosh, MD, MPH, Principal Investigator — Massachusetts Eye and Ear Infirmary; Claes H Dohlman, MD, PhD, Study Chair — Massachusetts Eye and Ear Infirmary; Mona Harissi-Dagher, MD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No